CLINICAL TRIAL: NCT03392883
Title: Scaling Up Science-based Mental Health Interventions in Latin America
Acronym: DIADA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Pontificia Universidad Javeriana (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lisa A. Marsch, Director of the Center for Technology and Behavioral Health, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1U19MH109988 D18019; 1U19MH109988 (NIH)
Record Dates: First submitted 2017-10-30; First posted 2018-01-08 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-10

CONDITIONS: Depression; Problematic Alcohol Use
Keywords: Latin America; Depression; mHealth; Problematic Alcohol Use
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The investigators will initially pilot test this mental health service delivery model at a single primary care site and then refine the model based on pilot data. The investigators will then expand implementation across 6 Colombia-based healthcare sites in urban and rural communities (including approximately 2000 participants). Consistent with a modified stepped wedge design (multiple baseline design), the investigators will implement the model across sites on a staggered basis and expand the number of sites in which the investigators implement over time. By conducting this multi-site implementation research project, the investigators can assess the extent to which the implementation model and associated outcomes are replicable across sites and/or the extent to which the model needs to be modified for differing contexts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Health Assisted Mental Healthcare (Experimental): This Digital Health Assisted Mental Healthcare intervention will be based on the novel mobile-based platform (Laddr® from Square2 Systems).
  Interventions: Behavioral: Laddr

INTERVENTIONS:
Behavioral: Laddr — Laddr is a mobile behavioral health technology that offers science-based self-regulation monitoring and health behavior change tools via an integrated platform to a wide array of populations. Specifically, the core functionality of Laddr (e.g., problem-solving therapy) will be structured to focus on an end user's management of depression and its impact on their functioning and quality of life. The program will secondarily focus on problematic alcohol use and its relationship to depression management.

SUMMARY:
Conduct systematic, multi-site mental health implementation research in both rural and urban primary care settings with a broad group of stakeholders in the US and Latin America.

DETAILED DESCRIPTION:
The investigators plan to launch and evaluate a new mental health service delivery model in Latin America. Specifically, in this new multi-component, mental health service delivery intervention, the investigators propose to: (1) harness mobile behavioral health technology for mental health (with a primary focus on depression and a secondary focus on problematic alcohol and other substance abuse), (2) launch new workforce training and service delivery models (including the integration of technology into service delivery), (3) launch and evolve an integrated data management system for systematic data tracking and outcomes assessment, and (4) launch and grow a learning collaborative of organizations integrating mental health into primary care. The investigators will launch this project at multiple primary care sites in various parts of Colombia, with a plan to inform subsequent adoption in several other Latin American countries, including Chile and Peru.

ELIGIBILITY:
Inclusion Criteria:

* Provider and administrative staff Inclusion Criteria:

  * Aged > 18 years
  * Have worked for the study site for at least 3 months.
* Participant Inclusion Criteria:

  * Aged > 18 years
  * Patients at one of our collaborating primary care sites
  * Screen positive for minor (score of 5-9), moderate (score of 10-14), moderately severe (score of 15-19) or severe (score of 20-27) depression on Patient Health Questionnaire (PHQ-9)62 and/or screen positive for problematic alcohol use on Alcohol Use Disorder Identification Test (AUDIT) developed by the World Health Organization (a score of 8 or more on 10-item AUDIT)63 and have a confirmed diagnosis of depression and/or alcohol use disorder based on clinical consultation at the primary care site
  * Willing to provide informed consent to use mobile intervention and complete study assessments

Exclusion Criteria:

-Participant Exclusion Criteria

* Diagnosis with co-occurring severe mental illness (e.g., schizophrenia, bipolar disorder, depression with psychotic features)
* Alcohol withdrawal symptoms that require higher level of care (e.g., emergency medical or inpatient treatment)
* Express suicidal intention. This assessment will be based on a combination of a patient's response on the PHQ-9 assessment followed by further assessment by a primary care clinician. The PHQ-9 measure will not be used solely to determine eligibility on this criterion. Persons who express suicidal intention will immediately be provided immediate crisis management in accordance with the crisis management protocol at the collaborating primary care site.
* Intoxicated or otherwise impaired at the time of assessment (rendering the individual incapable of informed consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1348 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Marsch, PhD, Principal Investigator — Dartmouth College; Carlos Gomez-Restrepo, MD, Principal Investigator — Pontificia Universidad Javeriana
Locations (6):
- Colombia (6):
  - ESE Hospital San Antonio de Guatavita, Guatavita, Cundinamarca
  - Hospital Mario Gaitán Yanguas, Soacha, Cundinamarca
  - Salud de Tundama, Duitama, Departamento de Boyacá
  - Empresa Social del Estado Hospital Regional de Duitama- Santa Rosa de Viterbo Branch, Santa Rosa de Viterbo, Departamento de Boyacá
  - Empresa Social del Estado Hospital Nelson Restrepo Martinez, Guayabal, Tolima Department
  - Javesalud, Bogotá

IPD SHARING:
Plan to Share IPD: Yes
The investigators agree to share all data in accordance with NIH's data sharing policy and in accordance with the specific data sharing requirements of this NIMH Cooperative Agreement funding mechanism. The investigators agree to cooperate with the NIMH program staff to provide timely, accurate, and complete data for purposes of monitoring the progress of research activities conducted within the proposed project. The investigators will also work with NIH program staff to promote broad availability of policies, practices, materials, tools and data generated by the proposed project activities. At the conclusion of this study, the investigators plan to make available a public use file of all related study data (stripped of all personal identifiers and suitable for use by other investigators). The investigators will make the dataset available in one or more several common formats (e.g., ascii tab delimited, SAS and SPSS).
Time Frame: Data will become available at the conclusion of the study. The investigators agree to retain records for each completed study for a minimum of 3 years (or more if necessary) after study data lock. The investigators will also comply with all relevant Institutional Review Board(s) IRB(s) and other regulatory entities regarding data sharing and records retention.
Access Criteria: Although the final dataset will be stripped of identifiers prior to release for sharing, the investigators will further assure participants' confidentiality with a data sharing agreement that stipulates that all data and associated documentation will only be available to users who declare: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. The investigators understand that NIH has access to any and all data generated under the cooperative agreement and agree to provide a royalty-free, nonexclusive, and irrevocable license for the government to reproduce, publish, or otherwise use the material and data derived from research conducted under this cooperative agreement.

REFERENCES:
- [Derived] Marsch LA, Gomez-Restrepo C, Bartels SM, Bell K, Camblor PM, Castro S, Cardenas Charry MP, Cepeda M, Cubillos L, John D, Jassir MP, Lemley SM, Suarez-Obando F, Torrey WC, Uribe JM, Williams MJ. Scaling Up Science-Based Care for Depression and Unhealthy Alcohol Use in Colombia: An Implementation Science Project. Psychiatr Serv. 2022 Feb 1;73(2):196-205. doi: 10.1176/appi.ps.202000041. Epub 2021 Aug 4. PMID 34347504

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the primary care site patients upon arrival were asked to complete screeners (for depression and problematic alcohol use). In the event of positive screen for depression and/or alcohol use problems, clinicians at site completed an in-depth diagnostic interview. Participants who met all inclusionary criteria were informed about this project and provided an informed consent form.
  Providers and administrators who worked for the site for at least 3 months were asked to participate.
Groups:
- Patients in Digital Health Assisted Mental Healthcare Intervention: Patients were offered a multi-component model of science-based mental health care. All participants who consented to participate were given access to the mobile therapeutic tool based on the novel mobile-based platform (Laddr® from Square2 Systems). A trained staff member at the primary care site showed them how to use the tool.
  Laddr is a mobile behavioral health technology that offers science-based self-regulation monitoring and health behavior change tools via an integrated platform to a wide array of populations. The program secondarily focused on problematic alcohol use and its relationship to depression management.
- Providers in Digital Health Assisted Mental Healthcare Intervention: Providers at partnering primary care sites were all offered the opportunity to complete the implementation context and outcome measure in this research project at the time of implementation launch and at designated timepoints thereafter.
- Administrative Staff in Digital Health Assisted Mental Healthcare Intervention: Administrative staff at partnering primary care sites were all offered the opportunity to complete the implementation context and outcome measure in this research project at the time of implementation launch and at designated timepoints thereafter.
Period: Overall Study
Arm/Group | Patients in Digital Health Assisted Mental Healthcare Intervention | Providers in Digital Health Assisted Mental Healthcare Intervention | Administrative Staff in Digital Health Assisted Mental Healthcare Intervention
Started | 1264 | 45 | 39
Completed | 928 | 32 | 30
Not Completed | 336 | 13 | 9
Not completed — Lost to Follow-up | 122 | 13 | 9
Not completed — Death | 4 | 0 | 0
Not completed — Lack of Efficacy | 29 | 0 | 0
Not completed — Withdrawal by Subject | 180 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Seventeen of the Baseline measures are not administered to providers and administrative staff. Therefore, there are zero participants analyzed among providers and administrative staff for those measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients in Digital Health Assisted Mental Healthcare Intervention | Providers in Digital Health Assisted Mental Healthcare Intervention | Administrative Staff in Digital Health Assisted Mental Healthcare Intervention | Total
Number analyzed (Participants) | 1264 | 45 | 39 | 1348
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.60 (17.28) | 32.87 (10.12) | 36.39 (12.51) | 48.88 (17.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 969 | 30 | 27 | 1026
  Male | 295 | 15 | 12 | 322
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 991 | 42 | 34 | 1067
  Not Hispanic or Latino | 20 | 0 | 1 | 21
  Unknown or Not Reported | 253 | 3 | 4 | 260
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 23 | 0 | 1 | 24
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 0 | 0 | 10
  White | 232 | 9 | 7 | 248
  More than one race | 681 | 22 | 23 | 726
  Unknown or Not Reported | 318 | 14 | 8 | 340
Region of Enrollment [Number; unit: participants]
  Colombia | 1264 | 45 | 39 | 1348
Name of Primary Care Center Site [Count of Participants; unit: Participants]
  Javesalud - Bogota | 483 | 13 | 12 | 508
  Hospital Regional de Duitama | 471 | 14 | 6 | 491
  Hospital Santa Rosa de Viterbo | 196 | 8 | 6 | 210
  Hospital Granja de Lerida | 27 | 5 | 9 | 41
  Hospital de Chaparral | 78 | 3 | 3 | 84
  Hospital Armero Guayabal | 9 | 2 | 3 | 14
  Prefer not to respond | 0 | 0 | 0 | 0
Education Level [Count of Participants; unit: Participants]
  None | 34 | 0 | 0 | 34
  Preschool | 1 | 0 | 0 | 1
  Kindergarten | 0 | 0 | 0 | 0
  Grade 1 | 64 | 0 | 0 | 64
  Grade 2 | 71 | 0 | 0 | 71
  Grade 3 | 72 | 0 | 0 | 72
  Grade 4 | 47 | 0 | 0 | 47
  Grade 5 | 178 | 0 | 0 | 178
  Grade 6 | 36 | 0 | 0 | 36
  Grade 7 | 43 | 0 | 0 | 43
  Grade 8 | 31 | 0 | 0 | 31
  Grade 9 | 40 | 0 | 0 | 40
  Grade 10 | 17 | 0 | 0 | 17
  Grade 11 | 21 | 0 | 0 | 21
  Secondary Education Diploma | 198 | 0 | 1 | 199
  Technical Studies | 149 | 2 | 9 | 160
  Less than one year of university | 18 | 0 | 1 | 19
  Diploma | 4 | 0 | 0 | 4
  University Degree | 8 | 2 | 1 | 11
  Master's Degree | 18 | 13 | 12 | 43
  Professional Degree | 135 | 28 | 14 | 177
  Doctorate | 1 | 0 | 0 | 1
  At least one year in two-year university program | 21 | 0 | 0 | 21
  One year in four-year university program | 13 | 0 | 0 | 13
  Two years in four-year university program | 9 | 0 | 0 | 9
  At least three years in four-year university program | 35 | 0 | 1 | 36
  Unknown or prefers not to respond | 0 | 0 | 0 | 0
Socioeconomic Status [Count of Participants; unit: Participants] — Socioeconomic stratification in Colombia is classified based on the residential neighborhood from 1-6, with 6 being the wealthiest and 1 the poorest. Official stratum in Colombia is found according to information on the participant's utility bill. Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Rural Area | 168 | 0 | 0 | 168
    Stratum 1 | 300 | 0 | 0 | 300
    Stratum 2 | 316 | 0 | 0 | 316
    Stratum 3 | 272 | 0 | 0 | 272
    Stratum 4 | 152 | 0 | 0 | 152
    Stratum 5 | 33 | 0 | 0 | 33
    Stratum 6 | 9 | 0 | 0 | 9
    Prefers not to respond | 14 | 0 | 0 | 14
Employment Status [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Full-time Employed | 171 | 0 | 0 | 171
    Self-employed | 286 | 0 | 0 | 286
    Part-time Employed | 49 | 0 | 0 | 49
    Unemployed, seeking jobs | 112 | 0 | 0 | 112
    Unemployed, not seeking jobs | 39 | 0 | 0 | 39
    Unable to work | 25 | 0 | 0 | 25
    Pensioner | 75 | 0 | 0 | 75
    Housekeeper | 428 | 0 | 0 | 428
    Student | 70 | 0 | 0 | 70
    Prefers not to respond | 9 | 0 | 0 | 9
Marital Status [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Single | 399 | 0 | 0 | 399
    Married or Free Union | 544 | 0 | 0 | 544
    Separated | 172 | 0 | 0 | 172
    Divorced | 36 | 0 | 0 | 36
    Widowed | 107 | 0 | 0 | 107
    Prefers not to respond | 6 | 0 | 0 | 6
Number of persons in household [Count of Participants; unit: Participants]
  0 | 130 | 0 | 0 | 130
  1 | 312 | 0 | 0 | 312
  2 | 277 | 0 | 0 | 277
  3 | 253 | 0 | 0 | 253
  4 | 148 | 0 | 0 | 148
  5 | 77 | 0 | 0 | 77
  6 | 33 | 0 | 0 | 33
  7 | 16 | 0 | 0 | 16
  8 | 8 | 0 | 0 | 8
  9 | 4 | 0 | 0 | 4
  10 | 1 | 0 | 0 | 1
  11 | 2 | 0 | 0 | 2
  12 | 1 | 0 | 0 | 1
  14 | 2 | 0 | 0 | 2
Health Insurance Status [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    No insurance | 1 | 0 | 0 | 1
    Subsidized plan (ARS, SISBEN, EPS-S) | 845 | 0 | 0 | 845
    Contributory plan (EPS) | 413 | 0 | 0 | 413
    Indigenous Health plan | 0 | 0 | 0 | 0
    Supplemental plan or prepaid medical plan | 4 | 0 | 0 | 4
    Special plan (Armed Forces, Ecopetrol) | 0 | 0 | 0 | 0
    Prefers not to respond | 1 | 0 | 0 | 1
Length of time to reach healthcare center [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    0-29 minutes | 631 | 0 | 0 | 631
    30-59 minutes | 464 | 0 | 0 | 464
    60-120 minutes | 134 | 0 | 0 | 134
    More than 120 minutes | 34 | 0 | 0 | 34
    Prefers not to respond | 1 | 0 | 0 | 1
History of previous depressive episodes [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    0 episodes | 890 | 0 | 0 | 890
    1 episode | 225 | 0 | 0 | 225
    2 episodes | 70 | 0 | 0 | 70
    3 episodes | 71 | 0 | 0 | 71
    Prefers not to respond | 8 | 0 | 0 | 8
History of Traumatic Events [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    No traumatic events | 500 | 0 | 0 | 500
    1 | 372 | 0 | 0 | 372
    2 | 199 | 0 | 0 | 199
    3 | 83 | 0 | 0 | 83
    4 | 37 | 0 | 0 | 37
    5 | 24 | 0 | 0 | 24
    6 | 10 | 0 | 0 | 10
    7 | 1 | 0 | 0 | 1
    9 | 1 | 0 | 0 | 1
    10 | 6 | 0 | 0 | 6
    Prefers not to respond | 31 | 0 | 0 | 31
Family History of Depression [Count of Participants; unit: Participants]
  Parents with depression | 163 | 0 | 0 | 163
  Siblings with depression | 133 | 0 | 0 | 133
  First degree relatives with depression | 132 | 0 | 0 | 132
  No family history of depression | 764 | 0 | 0 | 764
  Prefers not to respond | 156 | 0 | 0 | 156
Family History of Harmful Alcohol Use [Count of Participants; unit: Participants]
  Parents with harmful alcohol use | 473 | 0 | 0 | 473
  Siblings with harmful alcohol use | 356 | 0 | 0 | 356
  First degree relatives with harmful alcohol use | 367 | 0 | 0 | 367
  No family history of harmful alcohol use | 605 | 0 | 0 | 605
  Prefers not to respond | 18 | 0 | 0 | 18
Smartphone Use [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Yes - has a smartphone. | 882 | 0 | 0 | 882
    No - does not have a smartphone | 382 | 0 | 0 | 382
Internet Use [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Yes, uses the Internet | 843 | 0 | 0 | 843
    No, does not use the Internet | 421 | 0 | 0 | 421
Tobacco Use [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Current smoker | 163 | 0 | 0 | 163
    Former smoker | 414 | 0 | 0 | 414
    Never smoked | 686 | 0 | 0 | 686
    Prefers not to respond | 1 | 0 | 0 | 1
Antidepressants Use [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Yes | 187 | 0 | 0 | 187
    No | 1075 | 0 | 0 | 1075
    Prefers not to respond | 2 | 0 | 0 | 2
Psychotherapy Treatment Use [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Yes | 213 | 0 | 0 | 213
    No | 1048 | 0 | 0 | 1048
    Prefers not to respond | 3 | 0 | 0 | 3
Alcoholics Anonymous [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Yes | 12 | 0 | 0 | 12
    No | 1252 | 0 | 0 | 1252
    Prefers not to respond | 0 | 0 | 0 | 0
Medication for controlling problematic alcohol use [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Yes | 2 | 0 | 0 | 2
    No | 1262 | 0 | 0 | 1262
    Prefers not to respond | 0 | 0 | 0 | 0
Substance Use [Count of Participants; unit: Participants] — Population: This measure is not administered to providers and administrative staff.
  Participants
    Tobacco: number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Tobacco | 163 | 0 | 0 | 163
    Cannabis: number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Cannabis | 53 | 0 | 0 | 53
    Cocaine: number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Cocaine | 7 | 0 | 0 | 7
    Prescription Stimulants: number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Prescription Stimulants | 2 | 0 | 0 | 2
    Methamphetamine: number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Methamphetamine | 1 | 0 | 0 | 1
    Sedatives: number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Sedatives | 1 | 0 | 0 | 1
    Hallucinogens: number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Hallucinogens | 5 | 0 | 0 | 5
    Street Opioids: number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Street Opioids | 0 | 0 | 0 | 0
    Prescription Opioids: number analyzed (Participants) | 1264 | 0 | 0 | 1264
    Prescription Opioids | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Integrated Measure of Implementation Context and Outcomes as a Change Over Time in Low and Middle Income Countries Consumer Instrument
Description: This measure consists of 5 scales: Adoption, Appropriateness, Acceptability, Feasibility, and Reach/Access. All four scales have a range of 1 to 4 (1- Not at all, 2- A little bit, 3- A moderate amount, 4- A lot).
Time Frame: At 6- and 12-month follow-up visits with a sub-sample of participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients in Digital Health Assisted Mental Healthcare Intervention
Number analyzed (Participants) | 166
score on a scale
  6-month follow-up Adoption | 2.76 (0.58)
  6-month follow-up Acceptability | 3.22 (0.64)
  6-month follow-up Appropriateness | 3.21 (0.64)
  6-month follow-up Feasibility | 2.91 (0.62)
  6-month follow-up Reach/Access | 2.59 (0.69)
  12-month follow-up Adoption | 3.05 (0.62)
  12-month follow-up Acceptability | 3.27 (0.61)
  12-month follow-up Appropriateness | 3.28 (0.50)
  12-month follow-up Feasibility | 2.93 (0.54)
  12-month follow-up Reach/Access | 2.67 (0.66)
Statistical Analysis 1: Comparison: Patients in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time for every subscale. This Statistical Analysis describes the Adoption subscale results; Test type: Other — Paired version (T-test for paired sample, Friedman and McNemar tests) was used for contrasting the equality among the variables at different moments of time. In order to adjust our results by potential confounders, ANCOVA analyses was performed. Symmetric 95% confidence intervals will be provided for relevant parameters. All p-values were referred to two-sided hypotheses. P-values below 0.05 were considered statistically significant; p < 0.001, t-test, 2 sided — p<0.05 is the threshold for statistical significance
Statistical Analysis 2: Comparison: Patients in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time for every subscale in this instrument. This Statistical Analysis describes the Acceptability subscale results; Test type: Other; p = 0.552, t-test, 2 sided — p<0.05 is the threshold for statistical significance
Statistical Analysis 3: Comparison: Patients in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time for every subscale in this instrument. This Statistical Analysis describes the Appropriateness subscale results; Test type: Other; p = 0.320, t-test, 2 sided — p<0.05 is the threshold for statistical significance
Statistical Analysis 4: Comparison: Patients in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time for every subscale in this instrument. This Statistical Analysis describes the Feasibility subscale results; Test type: Other; p = 0.879, t-test, 2 sided — p<0.05 is the threshold for statistical significance
Statistical Analysis 5: Comparison: Patients in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time for every subscale in this instrument. This Statistical Analysis describes the Reach/Access subscale results; Test type: Other; p = 0.242, t-test, 2 sided — p<0.05 is the threshold for statistical significance

2. Primary Outcome: The Integrated Measure of Implementation Context and Outcomes as a Change Over Time in Low and Middle Income Countries Provider Instrument
Description: This measure consists of 8 scales: Adoption, Appropriateness, Feasibility, Reach/Access, Organizational climate, Leadership in Implementing, and General Leadership Skills. All eight scales have a range of 1 to 4 (1- Not at all, 2- A little bit, 3- A moderate amount, 4- A lot).
Time Frame: At the time of the provider training, 6 months, 12 months, 18 months, and 24 months.
Population: The study implementation timeline was designed to have staggered launch dates for the six sites. Specifically, Javesalud (Site 1) and Santa Rosa (Site 2) launched first and were able to complete all follow-ups. Tundama (Site 3) was only able to complete through 18-month follow-ups. Guasca (Site 4) and Armero (Site 5) were only able to complete through 12-month follow-ups. Soacha (Site 6) was only able to complete through the 6-month follow-ups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Providers in Digital Health Assisted Mental Healthcare Intervention
Number analyzed (Participants) | 24
score on a scale
  Adoption at Baseline | 2.95 (0.55)
  Adoption at 6 months: number analyzed (Participants) | 16
  Adoption at 6 months | 2.65 (0.61)
  Adoption at 12 months: number analyzed (Participants) | 22
  Adoption at 12 months | 2.93 (0.43)
  Adoption at 18 months | 2.92 (0.51)
  Adoption at 24 months: number analyzed (Participants) | 18
  Adoption at 24 months | 2.85 (0.68)
  Accessibility at Baseline | 3.41 (0.51)
  Accessibility at 6 months: number analyzed (Participants) | 16
  Accessibility at 6 months | 3.35 (0.45)
  Accessibility at 12 months: number analyzed (Participants) | 22
  Accessibility at 12 months | 3.50 (0.47)
  Accessibility at 18 months | 3.55 (0.32)
  Accessibility at 24 months: number analyzed (Participants) | 17
  Accessibility at 24 months | 3.38 (0.44)
  Appropriateness at Baseline | 3.40 (0.34)
  Appropriateness at 6 months: number analyzed (Participants) | 16
  Appropriateness at 6 months | 3.32 (0.47)
  Appropriateness at 12 months: number analyzed (Participants) | 22
  Appropriateness at 12 months | 3.52 (0.31)
  Appropriateness at 18 months | 3.41 (0.42)
  Appropriateness at 24 months: number analyzed (Participants) | 18
  Appropriateness at 24 months | 3.16 (0.48)
  Feasibility at Baseline | 2.94 (0.55)
  Feasibility at 6 months: number analyzed (Participants) | 16
  Feasibility at 6 months | 2.88 (0.38)
  Feasibility at 12 months: number analyzed (Participants) | 22
  Feasibility at 12 months | 2.72 (0.40)
  Feasibility at 18 months | 3.01 (0.31)
  Feasibility at 24 months: number analyzed (Participants) | 18
  Feasibility at 24 months | 2.84 (0.63)
  Resources at Baseline | 3.14 (0.65)
  Resources at 6 months: number analyzed (Participants) | 16
  Resources at 6 months | 3.08 (0.42)
  Resources at 12 months: number analyzed (Participants) | 22
  Resources at 12 months | 2.98 (0.47)
  Resources at 18 months | 3.17 (0.44)
  Resources at 24 months: number analyzed (Participants) | 18
  Resources at 24 months | 3.14 (0.64)
  Reach/Access at Baseline | 2.78 (0.65)
  Reach/Access at 6 months: number analyzed (Participants) | 16
  Reach/Access at 6 months | 2.85 (0.48)
  Reach/Access at 12 months: number analyzed (Participants) | 22
  Reach/Access at 12 months | 2.96 (0.44)
  Reach/Access at 18 months | 3.00 (0.52)
  Reach/Access at 24 months: number analyzed (Participants) | 18
  Reach/Access at 24 months | 2.91 (0.22)
  Organizational Climate at Baseline | 3.42 (0.44)
  Organizational Climate at 6 months: number analyzed (Participants) | 16
  Organizational Climate at 6 months | 3.43 (0.43)
  Organizational Climate at 12 months: number analyzed (Participants) | 22
  Organizational Climate at 12 months | 3.56 (0.30)
  Organizational Climate at 18 months | 3.60 (0.35)
  Organizational Climate at 24 months: number analyzed (Participants) | 18
  Organizational Climate at 24 months | 3.43 (0.61)
  Leadership in Implementing at Baseline | 3.38 (0.65)
  Leadership in Implementing at 6 months: number analyzed (Participants) | 16
  Leadership in Implementing at 6 months | 3.24 (0.64)
  Leadership in Implementing at 12 months: number analyzed (Participants) | 22
  Leadership in Implementing at 12 months | 3.46 (0.41)
  Leadership in Implementing at 18 months | 3.57 (0.44)
  Leadership in Implementing at 24 months: number analyzed (Participants) | 18
  Leadership in Implementing at 24 months | 3.06 (0.86)
  General Leadership Skills at Baseline | 3.32 (0.67)
  General Leadership Skills at 6 months: number analyzed (Participants) | 16
  General Leadership Skills at 6 months | 3.36 (0.55)
  General Leadership Skills at 12 months: number analyzed (Participants) | 22
  General Leadership Skills at 12 months | 3.48 (0.45)
  General Leadership Skills at 18 months | 3.48 (0.50)
  General Leadership Skills at 24 months: number analyzed (Participants) | 18
  General Leadership Skills at 24 months | 3.20 (0.94)
Statistical Analysis 1: Comparison: Providers in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time in this data for every sub-scale. This Statistical Analysis describes the Adoption subscale results; Test type: Other; p = 0.237, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 2: Comparison: Providers in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time in this data for every sub-scale. This Statistical Analysis describes the Accessibility subscale results; Test type: Other; p = 0.492, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 3: Comparison: Providers in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time in this data for every sub-scale. This Statistical Analysis describes the Appropriateness subscale results; Test type: Other; p = 0.285, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 4: Comparison: Providers in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time in this data for every sub-scale. This Statistical Analysis describes the Feasibility subscale results; Test type: Other; p = 0.964, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 5: Comparison: Providers in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time in this data for every sub-scale. This Statistical Analysis describes the Resources subscale results; Test type: Other; p = 0.942, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 6: Comparison: Providers in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time in this data for every sub-scale. This Statistical Analysis describes the Scope subscale results; Test type: Other; p = 0.366, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 7: Comparison: Providers in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time in this data for every sub-scale. This Statistical Analysis describes the Organizational Climate subscale results; Test type: Other; p = 0.021, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 8: Comparison: Providers in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time in this data for every sub-scale. This Statistical Analysis describes the Leadership in Implementing subscale results; Test type: Other; p = 0.832, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 9: Comparison: Providers in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time in this data for every sub-scale. This Statistical Analysis describes the General Leadership Skills subscale results; Test type: Other; p = 0.827, Regression, Linear — p<0.05 is the threshold for statistical significance

3. Primary Outcome: The Integrated Measure of Implementation Context and Outcomes as a Change Over Time in Low and Middle Income Countries Organizational Staff Instrument
Description: This measure consists of 9 scales: 1) Adoption, Appropriateness, Acceptability, Feasibility, Reach/Access, Organizational climate, Leadership in Implementing, General Leadership Skills, and Knowledge. All nine scales have a range of 1 to 4 (1- Not at all, 2- A little bit, 3- A moderate amount, 4- A lot).
Time Frame: At the time of the staff training, 6 months, 12 months, 18 months, and 24 months.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Administrative Staff in Digital Health Assisted Mental Healthcare Intervention: Administrative staff at partnering primary care sites will all be offered the opportunity to complete the implementation context and outcome measure in this research project at the time of implementation launch and at designated timepoints thereafter.
Arm/Group | Administrative Staff in Digital Health Assisted Mental Healthcare Intervention
Number analyzed (Participants) | 27
score on a scale
  Adoption at Baseline | 3.38 (0.47)
  Adoption at 6 months: number analyzed (Participants) | 20
  Adoption at 6 months | 3.37 (0.46)
  Adoption at 12 months: number analyzed (Participants) | 12
  Adoption at 12 months | 3.69 (0.40)
  Adoption at 18 months: number analyzed (Participants) | 21
  Adoption at 18 months | 3.87 (0.22)
  Adoption at 24 months: number analyzed (Participants) | 13
  Adoption at 24 months | 3.50 (0.67)
  Accessibility at Baseline | 3.77 (0.37)
  Accessibility at 6 months: number analyzed (Participants) | 20
  Accessibility at 6 months | 3.50 (0.39)
  Accessibility at 12 months: number analyzed (Participants) | 12
  Accessibility at 12 months | 3.50 (0.42)
  Accessibility at 18 months: number analyzed (Participants) | 21
  Accessibility at 18 months | 3.60 (0.42)
  Accessibility at 24 months: number analyzed (Participants) | 13
  Accessibility at 24 months | 3.39 (0.55)
  Appropriateness at Baseline | 3.54 (0.37)
  Appropriateness at 6 months: number analyzed (Participants) | 20
  Appropriateness at 6 months | 2.77 (0.89)
  Appropriateness at 12 months: number analyzed (Participants) | 12
  Appropriateness at 12 months | 2.99 (0.55)
  Appropriateness at 18 months: number analyzed (Participants) | 21
  Appropriateness at 18 months | 3.19 (0.53)
  Appropriateness at 24 months: number analyzed (Participants) | 13
  Appropriateness at 24 months | 3.07 (0.55)
  Feasibility at Baseline | 2.88 (0.60)
  Feasibility at 6 months: number analyzed (Participants) | 20
  Feasibility at 6 months | 3.17 (0.52)
  Feasibility at 12 months: number analyzed (Participants) | 12
  Feasibility at 12 months | 2.96 (0.55)
  Feasibility at 18 months: number analyzed (Participants) | 21
  Feasibility at 18 months | 3.20 (0.49)
  Feasibility at 24 months: number analyzed (Participants) | 13
  Feasibility at 24 months | 3.17 (0.59)
  Reach/Access at Baseline | 2.93 (0.58)
  Reach/Access at 6 months: number analyzed (Participants) | 20
  Reach/Access at 6 months | 3.41 (0.62)
  Reach/Access at 12 months: number analyzed (Participants) | 12
  Reach/Access at 12 months | 3.47 (0.54)
  Reach/Access at 18 months: number analyzed (Participants) | 21
  Reach/Access at 18 months | 3.70 (0.35)
  Reach/Access at 24 months: number analyzed (Participants) | 13
  Reach/Access at 24 months | 3.58 (0.27)
  Organizational Climate at Baseline | 3.39 (0.43)
  Organizational Climate at 6 months: number analyzed (Participants) | 20
  Organizational Climate at 6 months | 3.20 (0.77)
  Organizational Climate at 12 months: number analyzed (Participants) | 12
  Organizational Climate at 12 months | 3.22 (0.63)
  Organizational Climate at 18 months: number analyzed (Participants) | 21
  Organizational Climate at 18 months | 3.52 (0.64)
  Organizational Climate at 24 months: number analyzed (Participants) | 13
  Organizational Climate at 24 months | 3.47 (0.48)
  Leadership in Implementing at Baseline | 3.29 (0.69)
  Leadership in Implementing at 6 months: number analyzed (Participants) | 20
  Leadership in Implementing at 6 months | 3.17 (0.78)
  Leadership in Implementing at 12 months: number analyzed (Participants) | 12
  Leadership in Implementing at 12 months | 3.25 (0.80)
  Leadership in Implementing at 18 months: number analyzed (Participants) | 21
  Leadership in Implementing at 18 months | 3.65 (0.37)
  Leadership in Implementing at 24 months: number analyzed (Participants) | 13
  Leadership in Implementing at 24 months | 3.47 (0.45)
  General Leadership Skills at Baseline | 3.34 (0.56)
  General Leadership Skills at 6 months: number analyzed (Participants) | 20
  General Leadership Skills at 6 months | 2.42 (1.02)
  General Leadership Skills at 12 months: number analyzed (Participants) | 12
  General Leadership Skills at 12 months | 2.92 (0.81)
  General Leadership Skills at 18 months: number analyzed (Participants) | 21
  General Leadership Skills at 18 months | 2.44 (0.63)
  General Leadership Skills at 24 months: number analyzed (Participants) | 13
  General Leadership Skills at 24 months | 2.80 (1.05)
  Knowledge at Baseline | 1.95 (0.48)
  Knowledge at 6 months: number analyzed (Participants) | 20
  Knowledge at 6 months | 1.95 (0.28)
  Knowledge at 12 months: number analyzed (Participants) | 12
  Knowledge at 12 months | 1.92 (0.27)
  Knowledge at 18 months: number analyzed (Participants) | 21
  Knowledge at 18 months | 1.91 (0.26)
  Knowledge at 24 months: number analyzed (Participants) | 13
  Knowledge at 24 months | 1.92 (0.26)
Statistical Analysis 1: Comparison: Administrative Staff in Digital Health Assisted Mental Healthcare Intervention; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.118, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 2: Comparison: Administrative Staff in Digital Health Assisted Mental Healthcare Intervention; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.896, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 3: Comparison: Administrative Staff in Digital Health Assisted Mental Healthcare Intervention; [analysis description as in outcome 2, analysis 3]; Test type: Other; p = 0.739, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 4: Comparison: Administrative Staff in Digital Health Assisted Mental Healthcare Intervention; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = 0.724, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 5: Comparison: Administrative Staff in Digital Health Assisted Mental Healthcare Intervention; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.301, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 6: Comparison: Administrative Staff in Digital Health Assisted Mental Healthcare Intervention; [analysis description as in outcome 2, analysis 7]; Test type: Other; p = 0.034, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 7: Comparison: Administrative Staff in Digital Health Assisted Mental Healthcare Intervention; [analysis description as in outcome 2, analysis 8]; Test type: Other; p = 0.015, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 8: Comparison: Administrative Staff in Digital Health Assisted Mental Healthcare Intervention; [analysis description as in outcome 2, analysis 9]; Test type: Other; p = 0.081, Regression, Linear — p<0.05 is the threshold for statistical significance
Statistical Analysis 9: Comparison: Administrative Staff in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time in this data for every sub-scale. This Statistical Analysis describes the Knowledge subscale results; Test type: Other; p = 0.790, Regression, Linear — p<0.05 is the threshold for statistical significance

4. Primary Outcome: The Program Sustainability Assessment Tool (PSAT) Providers
Description: This instrument was developed from the Program Sustainability Assessment and consists of 7 scales: Environmental Support, Partnerships, Organizational Capacity, Program Evaluation, Program Adaptation, Communication with Public, and Communications within the organization. All scales have a range of 1 to 4 (1- Not at all, 2- A little bit, 3- A moderate amount, 4- A lot). The seven sub-scales are combined to an overall score by averaging the sub-scale scores. The computed overall scales have a range of 1 to 4.
Time Frame: At the time of the provider training, 6 months, 12 months, 18 months, and 24 months.
Population: The study implementation timeline was designed to have staggered launch dates for the six sites. For providers/staff, not all sites completed 18 and 24-month follow-up assessments. Also, baseline data is collected prior to site implementation launch. Some providers/administrators consented and provided data (at various follow-up times) after baseline implementation data collection took place at the sites.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Providers in Digital Health Assisted Mental Healthcare Intervention
Number analyzed (Participants) | 41
score on a scale
  Baseline overall | 3.01 (0.61)
  6 months follow-up overall: number analyzed (Participants) | 17
  6 months follow-up overall | 2.91 (0.63)
  12 months follow-up overall: number analyzed (Participants) | 18
  12 months follow-up overall | 2.99 (0.41)
  18 months follow-up overall: number analyzed (Participants) | 16
  18 months follow-up overall | 3.01 (0.51)
  24 months follow-up overall: number analyzed (Participants) | 9
  24 months follow-up overall | 2.82 (0.63)
Statistical Analysis 1: Comparison: Providers in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes in the overall scores over time; Test type: Other; p = 0.023, Regression, Linear — p<0.05 is the threshold for statistical significance

5. Primary Outcome: The Program Sustainability Assessment Tool (PSAT) Administrative Staff
Description: This instrument was developed from the Program Sustainability Assessment and consists of 7 scales: Environmental Support, Funding Stability, Partnerships, Organizational Capacity, Program Evaluation, Program Adaptation, Communication with Public, Communications within the organization, and Communication with Government. All seven scales have a range of 1 to 4 (1- Not at all, 2- A little bit, 3- A moderate amount, 4- A lot). The seven sub-scales are combined to an overall score by averaging the sub-scale scores. The computed overall scales have a range of 1 to 4.
Time Frame: At the time of the staff training, 6 months, 12 months, 18 months, and 24 months.
Population: The study implementation timeline was designed to have staggered launch dates for the six sites. For providers/staff, not all sites completed 18 and 24-month follow-up assessments. Also, baseline data was collected prior to site implementation launch. Some providers/administrators consented and provided data (at various follow-up times) after baseline implementation data collection took place at the sites.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Administrative Staff in Digital Health Assisted Mental Healthcare Intervention
Number analyzed (Participants) | 30
score on a scale
  Baseline overall | 2.72 (0.58)
  6 months follow-up overall: number analyzed (Participants) | 19
  6 months follow-up overall | 3.14 (0.37)
  12 months follow-up overall: number analyzed (Participants) | 14
  12 months follow-up overall | 3.23 (0.27)
  18 months follow-up overall: number analyzed (Participants) | 17
  18 months follow-up overall | 3.41 (0.29)
  24 months follow-up overall: number analyzed (Participants) | 6
  24 months follow-up overall | 3.32 (0.32)
Statistical Analysis 1: Comparison: Administrative Staff in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes in the overall scores over time in this data; Test type: Other; p = 0.589, Regression, Linear — p<0.05 is the threshold for statistical significance

6. Secondary Outcome: Patient Health Questionnaire (PHQ-8)
Description: A measure with 8 items used to assess depression. The total score of the scale ranges from 0 to 24, with 0 representing no significant depressive symptoms and 24 representing the most severe depressive symptoms.
Time Frame: This patient measure were assessed at baseline and every 3 months thereafter for a period of 12 months (for a total of 5 assessment timepoints per patient).
Population: Only patient participants with a depression diagnosis completed the PHQ assessment at all timepoints. The number of participants analyzed varies at each assessment timepoint due to participants unable to reach during the window of follow-up and participants who withdrew from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients in Digital Health Assisted Mental Healthcare Intervention
Number analyzed (Participants) | 1214
score on a scale
  Baseline | 11.32 (5.07)
  3-Month: number analyzed (Participants) | 990
  3-Month | 5.82 (5.09)
  6-Month: number analyzed (Participants) | 950
  6-Month | 5.51 (4.94)
  9-Month: number analyzed (Participants) | 902
  9-Month | 5.37 (4.67)
  12-Month: number analyzed (Participants) | 863
  12-Month | 4.67 (4.38)
Statistical Analysis 1: Comparison: Patients in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time by calculating the mean difference of the scores at baseline assessment and at 12-month follow-up assessment; Test type: Other; Mean Difference (Net) = -6.65

7. Secondary Outcome: 12-item World Health Organization Disability Assessment Schedule 2.0 (WHODAS)
Description: The WHODAS 2.0 assesses health-related difficulties across six different domains of functioning (cognition, mobility, self-care, socializing, life activities, and participation) that are linked conceptually and operationally to the International Classification of Functioning, Disability and Health (ICF). The scores assigned to 12 items are - "none" (1), "mild" (2) "moderate" (3), "severe" (4) and "extreme" (5). The scores for the 12 items are summed into a total score ranging from 12 (least severe) to 50 (most severe). The last 3 items of the assessment collect the number of days the reported health-related difficulties impact the participants in the past 90 days.
Time Frame: This patient measure were assessed at baseline and every 3 months for a period of 12 months (for a total of 5 assessment timepoints-level assessments per patient).
Population: The number of participants analyzed differs at each assessment timepoint due to a number of participants who were unable to reach during the designated window of assessment and participants who actively withdrew from the study for various non-safety related reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Patients in Digital Health Assisted Mental Healthcare Intervention: Patients were offered a multi-component model of science-based mental health care. All participants who consent to participate will be given access to the mobile therapeutic tool based on the novel mobile-based platform (Laddr® from Square2 Systems). A trained staff member at the primary care site will show them how to use the tool.
  Laddr is a mobile behavioral health technology that offers science-based self-regulation monitoring and health behavior change tools via an integrated platform to a wide array of populations. The program will secondarily focus on problematic alcohol use and its relationship to depression management.
Arm/Group | Patients in Digital Health Assisted Mental Healthcare Intervention
Number analyzed (Participants) | 1264
score on a scale
  Baseline Total Sum Score | 23.07 (7.72)
  3-Month Total Sum Score: number analyzed (Participants) | 1049
  3-Month Total Sum Score | 19.55 (7.30)
  6-Month Total Sum Score: number analyzed (Participants) | 999
  6-Month Total Sum Score | 19.32 (7.50)
  9-Month Total Sum Score: number analyzed (Participants) | 958
  9-Month Total Sum Score | 18.87 (6.98)
  12-Month Total Sum Score: number analyzed (Participants) | 928
  12-Month Total Sum Score | 18.59 (6.73)
Statistical Analysis 1: Comparison: Patients in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time by calculating the mean difference of the total scores (sum of 12 items) at baseline assessment and at 12-month follow-up assessment; Test type: Other; Mean Difference (Net) = -4.48

8. Secondary Outcome: General Anxiety Disorder Screener (GAD-7)
Description: The GAD-7 is a 7-item self-reported screening questionnaire that has been validated to assess for generalized anxiety disorder (GAD) in outpatient and primary care settings. The measure is scored from 0 to 21, with 0 meaning minimal anxiety and 21 meaning most severe anxiety.
Time Frame: This patient measure were assessed at baseline and every 3 months for a period of 12 months (for a total of 5 assessment timepoints per patient).
Population: Number of participants analyzed differ at each assessment timepoint because some participants were unable to be reached during the designated window of follow-up and some participants withdrew from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients in Digital Health Assisted Mental Healthcare Intervention
Number analyzed (Participants) | 1264
score on a scale
  Baseline | 9.11 (5.43)
  3-Month: number analyzed (Participants) | 1021
  3-Month | 5.21 (4.65)
  6-Month: number analyzed (Participants) | 977
  6-Month | 4.63 (4.35)
  9-Month: number analyzed (Participants) | 933
  9-Month | 4.05 (3.97)
  12-Month: number analyzed (Participants) | 897
  12-Month | 3.34 (3.69)
Statistical Analysis 1: Comparison: Patients in Digital Health Assisted Mental Healthcare Intervention; [analysis description as in outcome 6, analysis 1]; Test type: Other; Mean Difference (Net) = -5.77

9. Secondary Outcome: The Quick Drinking Screen (QDS) (for Full Implementation Study Only)
Description: The Quick Drinking Screen (QDS) is a 3-item questionnaire which asks about average drinking habits over the last ninety days. The responses are used to calculate the number of standard drinks consumed per week. In this measure, a standard drink is defined as 1-12 oz. regular can or glass of beer, or 1-5 oz. glass of regular wine, or 1 ½ oz. of regular proof hard liquor or spirits. Patients with alcohol use disorder will be asked to complete this measure as part of the baseline assessment and at every 3 months follow-up (a total of 5 assessment timepoints).
Time Frame: At baseline and every 3 months for a period of 12 months (for a total of 5 assessment timepoints per patient with implementation study participants).
Population: The overall number of participants is different from the overall number of the patients arm, because this assessment was only administered to patients diagnosed with alcohol use disorder. There are different numbers of participants analyzed at each timepoint due to a number of participants who were unable to be reached in the designated window of follow-up and who withdrew from the study.
Measure: Mean (Standard Deviation); unit: standard drinks per week
Arm/Group | Patients in Digital Health Assisted Mental Healthcare Intervention
Number analyzed (Participants) | 168
standard drinks per week
  Baseline Standard Drinks per Week | 22.74 (28.28)
  3-Month Standard Drinks per Week: number analyzed (Participants) | 130
  3-Month Standard Drinks per Week | 35.20 (96.14)
  6-Month Standard Drinks per Week: number analyzed (Participants) | 115
  6-Month Standard Drinks per Week | 46.37 (102.00)
  9-Month Standard Drinks per Week: number analyzed (Participants) | 108
  9-Month Standard Drinks per Week | 38.11 (80.02)
  12-Month Standard Drinks per Week: number analyzed (Participants) | 105
  12-Month Standard Drinks per Week | 25.33 (72.61)
Statistical Analysis 1: Comparison: Patients in Digital Health Assisted Mental Healthcare Intervention; We analyzed changes over time by calculating the mean difference of the number of standard drinks per week at baseline assessment and at 12-month follow-up assessment; Test type: Other; Mean Difference (Net) = -2.59

10. Other Pre Specified Outcome: EuroQOL Five Dimensions Questionnaire (EQ-5D) (Only for Pilot Participants)
Description: The EQ-5D. The EQ-5D is a standardized instrument that has been widely used and validated within Spanish speaking populations from several countries in Latin America, and assesses 5 key dimensions of health.
Time Frame: This patient measure will be assessed at baseline and every 3 months for a period of 12 months (for a total of 5 assessment timepoints per patient with pilot participants).
Reporting Status: Not Posted

11. Other Pre Specified Outcome: EuroQol Visual Analogue Scale (EQ-VAS) (Only for Pilot Participants)
Description: The EQ-VAS assess health-related quality of life. The EQ-VAS asks "how good or bad your health is today?" The scale ranges from 0 (worst health imaginable) to 100 (best health imaginable). The participants marks their number with an "X" on the scale and writes it in a box.
Time Frame: as for outcome 10
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Alcohol Timeline Follow-back (Alcohol TLFB) (Only for Pilot Participants)
Description: A measure used to assess problematic alcohol use. The Alcohol TLFB asks patients about their alcohol use in the past 30 days.
Time Frame: as for outcome 10
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Behavioral Health Integration in Medical Care Index (BHIMC)
Description: The BHIMC is an organizational measure of the level of behavioral health integration in medical practice settings. It evaluates policy, clinical practice and workforce dimensions of integration using mixed methods, i.e. combination of document review and observation.
Time Frame: Approximately every year prior to the time of implementation launch at a given site (starting with baseline in late 2017); at the time of implementation launch; and approximately every year thereafter at each site until study completion (April 2021).
Reporting Status: Not Posted

14. Other Pre Specified Outcome: The Time-driven Activity-based Costing (TDABC) Approach
Description: The TDABC method measures costs of implementing the proposed model of care for depression and alcohol use disorders.The TDABC method will be used to determine the costs of the specific human, equipment, and facility resources used for delivering mental health care to patients as part of the model of care.
Time Frame: as for outcome 13
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Non-Study Medical and Other Services (NSMOS)
Description: The NSOMS assesses patients' medical resource use that is not part of the intervention, including non-treatment therapy visits, physician visits, residential and/or hospital detoxification, hospital and emergency department visits, and medication use through patient self-report.
Time Frame: At baseline and every 3 months for a period of 12 months (for a total of 5 assessment timepoints per patient).
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Non-Medical Expenses for Depression (NMED)
Description: The NMED assesses the non-medical costs of depression. This measure is in Spanish and has been used in Latin America and used by our team at Javeriana.
Time Frame: At baseline and every 3 months for a period of 12 months (for a total of 5 assessment timepoints per patient).
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Health and Work Performance Questionnaire (HPQ)
Description: The HPQ was developed by the World Health Organization, and assess the impact of depression on work performance (including sickness absence, presenteeism, and critical incidents).
Time Frame: At baseline, 6-month follow-ups, and 12-month follow-ups (for a total of 3 assessment timepoints per patient).
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Administrative Interviews
Description: Administrative interviews will assess implementation experiences, challenges to implementation and strategies used to facilitate implementation with different patient populations, changes made to workflow with use of the intervention, and salience of monitoring and feedback processes to inform providers and other stakeholders about the implementation success (approx. 5 at each site). The investigators will also assess the extent to which patients initiated use of the program via inquiry of their providers after learning of the program through patient channels.
Time Frame: At 3- and 6-months post-implementation (+/- a 2 week window around the targeted data collection date)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Patient Utilization Interviews/Observations
Description: The investigators will recruit and follow a sample of patients (approx. 5 at each site) during the implementation project to explore feasibility issues regarding use, barriers and facilitating strategies for using the program, optimal dissemination strategies for promoting use of the program, and overall experiences using the program over time. These patient participants will be encouraged to document their experiences with the mental health service delivery model in an ongoing manner (e.g., note jotting, pictures, audio recording).
Time Frame: At 3- and 6-months post-implementation (+/- a 2 week window around the targeted data collection date)
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Provider Interviews
Description: Provider interviews will assess implementation experiences, challenges to implementation and strategies used to facilitate implementation with different patient populations, changes made to workflow with use of the intervention, and salience of monitoring and feedback processes to inform providers and other stakeholders about the implementation success (approx. 5 at each site). The investigators will also assess the extent to which patients initiated use of the program via inquiry of their providers after learning of the program through patient channels.
Time Frame: At 3- and 6-months post-implementation (+/- a 2 week window around the targeted data collection date)
Reporting Status: Not Posted

21. Other Pre Specified Outcome: COVID-19 Impact Survey
Description: The COVID-19 Impact Survey is a self-reported questionnaire developed by the NIMH U19 Scale-Up Hubs and will assess the impact of COVID-19 among patients, providers, and administrators enrolled in this study. Given the unknown and widespread implications of the COVID-19 pandemic in Colombia, it is critical to understand the context of COVID-19 for interpreting the study's findings.
Time Frame: Patients will be assessed once at a follow-up visit every 3 months or at a separately scheduled visit. Providers and administrators will be assessed once at a follow-up visit every 6 months or at a separate visit.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months after baseline assessment.
Description: The study collected and reported adverse events only for patient participants. Adverse event collection was not conducted for providers and administrators.
Groups:
- Patients in Digital Health Assisted Mental Healthcare Intervention: Patients will be offered a multi-component model of science-based mental health care. All participants who consent to participate will be given access to the mobile therapeutic tool based on the novel mobile-based platform (Laddr® from Square2 Systems). A trained staff member at the primary care site will show them how to use the tool.
  Laddr is a mobile behavioral health technology that offers science-based self-regulation monitoring and health behavior change tools via an integrated platform to a wide array of populations. The program will secondarily focus on problematic alcohol use and its relationship to depression management.
Arm/Group | Patients in Digital Health Assisted Mental Healthcare Intervention
All-Cause Mortality (participants affected / at risk) | 7/1264
Serious Adverse Events (participants affected / at risk) | 107/1264
Other Adverse Events (participants affected / at risk) | 615/1264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients in Digital Health Assisted Mental Healthcare Intervention (N=1264)
Suicidality (Psychiatric disorders) | 28
Paralysis due to Parkinson's Disease (Nervous system disorders) | 1
Hospitalization due to Diarrhea (Gastrointestinal disorders) | 1
Chest Pain (Cardiac disorders) | 5
Hospitalization due to Hyperglycemia (Blood and lymphatic system disorders) | 1
Spinal Surgery (Surgical and medical procedures) | 1
Heart Dysfunction (Cardiac disorders) | 8
Thyroidectomy (Endocrine disorders) | 1
Removal of Gallbladder (Gastrointestinal disorders) | 4
Catheterization (Surgical and medical procedures) | 2
Liver Complications (Gastrointestinal disorders) | 1
Renal Procedure (Renal and urinary disorders) | 2
Broken Limb (Injury, poisoning and procedural complications) | 4
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Colon Procedure (Surgical and medical procedures) | 1
Breast Cancer Related Surgery and Treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Shingles (Infections and infestations) | 1
Manic Episode (Psychiatric disorders) | 1
Total Knee Replacement (Surgical and medical procedures) | 1
Caesarean Section Procedure (Surgical and medical procedures) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Epilepsy (Nervous system disorders) | 3
Urinary Tract Infection (Infections and infestations) | 3
Infection in Leg (Infections and infestations) | 1
Facial Paralysis (Nervous system disorders) | 3
Curettage Biopsy (Surgical and medical procedures) | 1
Hernia Repair (Surgical and medical procedures) | 3
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Worsening Depression without Suicidality (Psychiatric disorders) | 3
Surgery for Hand Trauma (Surgical and medical procedures) | 1
Blood Transfusion for Anemia (Blood and lymphatic system disorders) | 1
Cysts (General disorders) | 1
Hip Replacement (Surgical and medical procedures) | 1
Endoscopic retrograde cholangiopancreatography (Surgical and medical procedures) | 1
Hospitalization due to COVID-19 Infection (Infections and infestations) | 21
Herniated Disc (Musculoskeletal and connective tissue disorders) | 1
Arthroscopy Procedure (Surgical and medical procedures) | 1
Appendectomy (Surgical and medical procedures) | 1
Gastritis (General disorders) | 1
Abdominal Pain (Surgical and medical procedures) | 1 — Hospitalization for related tests and scans
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients in Digital Health Assisted Mental Healthcare Intervention (N=1264)
Medical appointment due to non-serious diagnosis related symptoms (Psychiatric disorders) | 403
COVID-19 Infection (Infections and infestations) | 84
Headaches (General disorders) | 4
Vertigo Episode (Nervous system disorders) | 2
Resection of Malignant Mass on Face (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Displacement and imbalance (Nervous system disorders) | 1
Facial Paralysis (Nervous system disorders) | 1
Fever and face rash (General disorders) | 1
Complication of chronic venous insufficiency (Blood and lymphatic system disorders) | 1
Worsening of Depressive Symptoms (Psychiatric disorders) | 23
Panic attack (Psychiatric disorders) | 10
Suicide ideation with risk of self-harm (Psychiatric disorders) | 7
Worsening of depression symptoms secondary to autoimmune disease complication (Psychiatric disorders) | 1
Parasuicide behavior (Psychiatric disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 11
Excision of Uterine Fibroid (Reproductive system and breast disorders) | 2
Tubal ligation surgery (Reproductive system and breast disorders) | 1
Ovary and thyroid cysts (Reproductive system and breast disorders) | 1
Excision of ovarian myoma (Reproductive system and breast disorders) | 1
Post-abortion difficulties (Reproductive system and breast disorders) | 1
Pregnancy miscarriage (Pregnancy, puerperium and perinatal conditions) | 1
Bleeding related to pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Vaginal bleeding (Reproductive system and breast disorders) | 1
Resection of endometrial polyps (Reproductive system and breast disorders) | 1
Trauma related to fall injuries (Injury, poisoning and procedural complications) | 7
Work accident (Injury, poisoning and procedural complications) | 2
Accident under alcohol influence (Injury, poisoning and procedural complications) | 1
Eye Procedure (Eye disorders) | 5
Ocular hemorrhage (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Food poisoning (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Resection of Gastric and Duodenal Polyps (Gastrointestinal disorders) | 1
Stomach virus (Gastrointestinal disorders) | 1
Liquid stools (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Respiratory problems (Respiratory, thoracic and mediastinal disorders) | 3
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Chest pain (Cardiac disorders) | 3
Pacemaker procedure (Cardiac disorders) | 1
Arrythmia Tachycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Varicose Vein Surgery (Cardiac disorders) | 1
Heart murmur (Cardiac disorders) | 1
Ankle trauma (Injury, poisoning and procedural complications) | 2
Mild Carpal Tunnel (Musculoskeletal and connective tissue disorders) | 1
Hyperextension in Spine (Musculoskeletal and connective tissue disorders) | 1
Broken Finger (Musculoskeletal and connective tissue disorders) | 1
Spinal surgery (Musculoskeletal and connective tissue disorders) | 1
Broken arm (Musculoskeletal and connective tissue disorders) | 1
Knee pain (Musculoskeletal and connective tissue disorders) | 1
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1
Vocal cords surgery (Musculoskeletal and connective tissue disorders) | 1
Diabetes diagnosis (Renal and urinary disorders) | 1
Kidney stone (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Tiroidectomy (Endocrine disorders) | 1
Biopsy of thyroid nodules (Endocrine disorders) | 1

LIMITATIONS AND CAVEATS:
On March 23, 2020, our study staff paused participant recruitment and all face-to-face activities at all of our study's sites due to COVID-19 related safety concerns. The study has not recruited patient participants since that date. On May 15, 2020, the study implemented a remote consent process to allow study enrollment of eligible providers and administrators and a remote informed consent process to allow all participants to participate in the qualitative sub-study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT03392883/Prot_SAP_002.pdf
  • Informed Consent Form: Patient Informed Consent form (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT03392883/ICF_000.pdf
  • Informed Consent Form: Staff Informed Consent form (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT03392883/ICF_001.pdf